CLINICAL TRIAL: NCT05117658
Title: A Single-Arm, Multi-Centre, Open-Label Phase II Study of HA121-28 in Patients With RET Fusion-Positive Advanced Non-Small Cell Lung Cancer
Brief Title: Study of HA121-28 in Patients With Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HA122-CSP-004
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2021-12

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HA121-28 (Experimental): Patients will receive HA121-28 tablets at 450 mg once daily (QD) for 21 days on a 28-day treatment cycle.
  Interventions: Drug: HA121-28 tablet

INTERVENTIONS:
Drug: HA121-28 tablet — HA121-28 tablet, 450 mg, po, QD×21 days, every 4 weeks (28 days)

SUMMARY:
This study is a multicenter, open-label, single-arm phase II study to evaluate efficacy and safety of HA121-28 tablets in patients with rearranged during transfection (RET) fusion-positive advanced non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this study and sign the informed consent form;
2. Aged 18 ~ 75 years old (inclusive), male or female;
3. Patients with histologically or cytologically confirmed unresectable locally advanced or metastatic non-small cell lung cancer;
4. RET gene fusion, as demonstrated by "Next-generation" sequencing(NGS) method in central laboratory with College of American Pathologists(CAP) or Clinical Laboratory Improvement Amendments(CLIA) certification;
5. Progressive disease after at least one line of standard therapy (including patients with disease progression during or within 6 months of the end of adjuvant therapy);
6. At least one measurable lesion according to RECIST 1.1 (for lesions previously treated with radiation, the lesion can be included as a measurable lesion only if there is clear disease progression after radiotherapy);
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score 0-1;
8. Adequate organ function, laboratory tests meeting the following criteria:

   * Neutrophil count (ANC) ≥ 1.5 × 10^9/L (no G-CSF for WBC-elevating therapy within 2 weeks prior to the laboratory test);
   * Platelet count (PLT) ≥ 75 × 10^9/L (no platelet transfusion or other drugs to promote platelet production within 2 weeks prior to the laboratory test);
   * Hemoglobin (Hb) ≥ 90 g/L; (not receiving red blood cell transfusion or erythropoiesis-stimulating drugs within 2 weeks prior to the laboratory test);
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × upper limit of normal (ULN) (≤ 5.0 × ULN for patients with liver metastases);
   * Serum total bilirubin (TBIL) ≤ 1.5 × ULN;
   * Serum creatinine ≤ 1.5 × ULN;
   * Albumin ≥ 30 g/L;
9. Male and female patients of childbearing age agree to take effective contraceptive measures during treatment and within 6 months after the completion of treatment.

Exclusion Criteria:

1. Had a documented oncogenic driver gene alteration other than RET in NSCLC, ie, activating EGFR, BRAF, or KRAS mutation, MET exon 14 skipping mutation or high-level amplification, and ALK, ROS1, or NTRK1/2/3 gene fusions;
2. Prior treatment with selective RET inhibitors (including investigational selective RET inhibitors, such as LOXO-292, BLU-667, RXDX-105, etc.);
3. Patients who previously received any anti-tumor therapy (including but not limited to chemotherapy, radiotherapy and targeted therapy, etc.) within 4 weeks before the first use of the study drug; traditional Chinese medicine or Chinese patent medicine with anti-tumor indications within 2 weeks; local palliative radiotherapy for the relief of bone metastasis pain within 2 weeks;
4. Abnormal coagulation function (INR > 1.5 or APTT > 1.5 × ULN); patients with bleeding tendency (such as active peptic ulcer) or receiving thrombolytic or anticoagulant therapy;
5. Urine routine showed urine protein ≥ + + and 24 h urine protein > 1.0 g;
6. Patients who have undergone major surgical procedures within 4 weeks before the first dose or are expected to undergo major surgery during the study;
7. Patients with central nervous system (CNS) metastases who present with progressive neurological symptoms or require an increase in corticosteroid dose to control their CNS disease. If a patient requires treatment with corticosteroids for CNS disease, the dose must be stable for two weeks prior to the first dose;
8. Presence of poorly controlled pericardial, pleural, or peritoneal effusion;
9. Interstitial pneumonia requiring steroid therapy, drug-induced pneumonitis, radiation pneumonitis (except for stable radiation pneumonitis);
10. Significant cardiovascular disease, such as heart failure greater than New York Heart Association (NYHA) Class 2, unstable angina, serious arrhythmia, myocardial infarction or stroke within 6 months prior to the first dose, poorly controlled hypertension (defined as systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg on multiple measurements while on medication);
11. Patients who met any of the following criteria will be excluded:

    * QT interval (QTcF) value ≥ 470 ms for females and ≥ 450 ms for males; or congenital long QT syndrome, taking drugs known to prolong QT interval, family history of long QT syndrome;
    * Resting ECG showed any clinically significant abnormalities in rhythm, conduction, or morphology that required clinical intervention;
    * Cardiac ejection fraction less than 50%;
12. Patients with active hepatitis B virus or hepatitis C virus infection:

    * HBsAg positive with HBV DNA higher than the upper limit of normal range of the study site;
    * HCV antibody positive with HCV RNA higher than upper limit of normal range of the site;
13. Human immunodeficiency virus infected (HIV positive);
14. Inability or severe dysphagia;
15. Patients who have suffered from or are complicated with any other malignant tumor within 5 years (except radically resected skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, local prostate cancer, in situ cervical cancer or other carcinoma in situ);
16. Presence of any severe and/or uncontrolled disease that may affect the drug evaluation in the judgment of the investigator, including but not limited to: life-threatening autoimmune system diseases; drug abuse; severe nervous system diseases (such as epilepsy, dementia, etc.); history of severe mental disorders; severe infection, etc.;
17. Pregnant or lactating women;
18. Other conditions that, in the opinion of the investigator, make participation in the study unsuitable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 12 months
  The percentage of patients who achieve a complete response (CR) or partial response (PR) evaluated by Independent Review Committee (IRC) according to RECIST 1.1.

SECONDARY OUTCOMES:
ORR | Up to approximately 12 months
  The percentage of patients who achieve a CR or PR evaluated by investigator according to RECIST 1.1.
Progression-Free Survival (PFS) | Up to approximately 12 months
  Time from date of the first dose to date of recorded disease progression or death, whichever occurs first.
PFS | Up to approximately 12 months
  Evaluated by investigator.
Overall survival (OS) | Up to approximately 24 months
  Time from date of the first dose to date of death from any cause.
Disease Control Rate (DCR) | Up to approximately 12 months
  The percentage of patients who achieve a CR, PR or stable disease (SD) evaluated by IRC.
DCR | Up to approximately 12 months
  Evaluated by investigator.
Duration of Response (DOR) | Up to approximately 12 months
  Time from first documented response (CR or PR, whichever occurs first, evaluated by IRC) to date of disease progression or death due to any cause, whichever occurs first.
DOR | Up to approximately 12 months
  Evaluated by investigator.
Incidence of treatment-related adverse events (AEs) and serious adverse events (SAEs). | Up to 28 days after the last administration of HA121-28
  The AEs and SAEs will be assessed according to the National Cancer Institute (NCI) CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Centre, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Ruan DY, Huang WW, Li Y, Zhao Y, Shi Y, Jia Y, Cang S, Zhang W, Shi J, Chen J, Lin J, Liu Y, Xu J, Ouyang W, Fang J, Zhuang W, Liu C, Bu Q, Li M, Meng X, Sun M, Yang N, Dong X, Pan Y, Li X, Qu X, Zhang T, Yuan X, Hu S, Guo W, Li Y, Li S, Liu D, Song F, Tan L, Yu Y, Yu X, Zang A, Sun C, Zhang Q, Zou K, Dan M, Xu RH, Zhao H. Safety, pharmacokinetics and efficacy of HA121-28 in patients with advanced solid tumors and RET fusion-positive non-small-cell lung cancer: a multicenter, open-label, single-arm phase 1/2 trial. Signal Transduct Target Ther. 2025 Feb 28;10(1):62. doi: 10.1038/s41392-025-02155-5. PMID 40016191